CLINICAL TRIAL: NCT07107386
Title: An Observational, Longitudinal Study to Characterize the Dynamic Structure of Molecular and Digital Health Data in Healthy Older Adults
Brief Title: Temporal Investigation of Multimodal Elements
Acronym: TIME
Status: Recruiting | Type: Observational
Sponsor: Buck Institute for Research on Aging (Other)
Collaborators: Phenome Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: BUCK 2502; 1AY2AX000072-01 (Other Grant/Funding Number: ARPA-H)
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The TIME Study is a research project aiming to understand the body's natural rhythms. The goal is to see how daily and weekly changes in our bodies-from what's happening at a molecular level to data from wearable devices-are connected.

What is the study about? This study is trying to create a detailed map of how a person's body changes over time. By looking at information from blood, urine, and other samples, as well as data from smartwatches and other devices, researchers want to learn how our bodies' natural cycles work in healthy older adults. The long-term goal is to use this knowledge to help develop more personalized healthcare in the future.

Who can participate? The study is looking for healthy adults, age 55 or older, who have a smartphone and are able to travel to the Buck Institute in Novato, California, for study visits.

Participants will be asked to:

Attend weekly visits over 11 weeks to provide blood and other samples.

Wear health-tracking devices like a smart ring and watch.

Use a smartphone app to answer questions about their daily routines.

Complete two "challenge" tests, including drinking a glucose solution and exercising on a stationary bicycle.

Return for follow-up visits after 6 and 12 months.

Are there any risks or benefits? Benefits: There are no direct health benefits for participants. However, the information gained will help scientists create better diagnostic tools and treatments for future generations.

Risks: The main risks are minor discomfort from things like blood draws or skin irritation from the wearable devices. All personal information and data are kept private and secure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 55 years or older.
* Own a smartphone capable of running study-specific apps.
* Willing and able to attend in-person visits at the Buck Institute in Novato, CA.
* Reside in the Pacific or Mountain Time Zones.
* Able to speak, read, and write English.
* Willing to wear study devices continuously and allow researchers access to all data.
* Able to provide informed consent.

Exclusion Criteria:

* Hospitalization within the last 3 months.
* Needing assistance with daily living activities.
* Working night or irregular shifts.
* Certain musculoskeletal, pulmonary, or cardiovascular conditions.
* Uncontrolled high blood pressure (BP > 180/100 mmHg).
* Bleeding disorders, anemia requiring treatment, or recent blood donation.
* Poor vein access.
* Unstable health conditions.
* Chronic antibiotic use.
* Certain psychiatric disorders.
* Use of excluded medications, supplements, or products, including certain antibiotics or frequent sleep aids.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy older adults aged 55 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Generation of a longitudinal multi-omic and digital health dataset characterizing biorhythms in older adults | 12 months
  Establish a publicly shareable reference dataset integrating blood-based proteomic, metabolomic, and lipidomic profiles with continuous digital health data and microbiome samples from healthy older adults over time, capturing daily, weekly, and perturbation-induced physiological dynamics.

SECONDARY OUTCOMES:
Characterization of associations between molecular biomarkers and digital health data across time | 12 months
  Identify and quantify temporal correlations between blood-derived molecular biomarkers and physiological signals collected via wearable devices, including responses to standardized challenges.

CONTACTS AND LOCATIONS:
Overall Officials: James Yurkovich, PhD, Principal Investigator — Phenome Health, The Buck Institute for Research on Aging
Locations (1):
- Buck Institute, Novato, California, United States

IPD SHARING:
Plan to Share IPD: Undecided